CLINICAL TRIAL: NCT00396240
Title: ORBITAL: Open-Label Primary Care Study: Rosuvastatin Based Compliance Initiatives Linked To Achievement Of LDL Goals
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: study cancelled prior to FSI
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3560L00008; ORBITAL
Record Dates: First submitted 2006-11-03; First posted 2006-11-06 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Primary Hypercholesterolaemia
Keywords: rosuvastatin; hypercholesterolaemia; cholesterol; LDL-C; triglyceride; plasma lipids; compliance
MeSH Terms: conditions — Hypercholesterolemia; Patient Compliance | interventions — Rosuvastatin Calcium

INTERVENTIONS:
Drug: Rosuvastatin
Procedure: Initiatives to improve compliance

SUMMARY:
24 week open label study to compare the treatment either with rosuvastatin or rosuvastatin plus initiatives to improve compliance. If the subject does not reach the EAS LDL-C treatment goal at week 12, rosuvastatin will be titrated from 10mg to 20mg.

ELIGIBILITY:
Inclusion Criteria:

* Primary hypercholesterolaemia:
* Statin naïve subjects (LDL-C level > 3.5 mmol/L) or subjects on an ineffective "start dose" of a lipid-lowering therapy (LDL-C level > 3.1 mmol/L).
* CV risk > 20%,
* history of CHD or other established atherosclerotic disease

Exclusion Criteria:

* History of severe adverse events with another HMG-CoA reductase inhibitor
* Secondary hypercholesterolaemia;
* Unstable cardiovascular disease;
* Uncontrolled diabetes, active liver disease;
* Severe hepatic or renal impairment;
* Treatment with cyclosporin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1294
Dates: Start 2002-02

PRIMARY OUTCOMES:
Comparison of the rosuvastatin therapy (10mg daily, titrated to 20mg at 12 weeks if necessary), alone or in combination with enhanced compliance initiatives, at 6 months, in bringing subjects with prim. hypercholesterolaemia to the EAS LDL-C target goals

SECONDARY OUTCOMES:
To investigate the effect of rosuvastatin, both with and without compliance initiatives on number and percentage of subjects within the EAS or local LDL-C and TC target goals after 12 week therapy,
Safety of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Billeter, MD, Study Director — AstraZeneca; W. Riesen, MD, Principal Investigator — Cantonal Hospital of St. Gallen; R. Darioli, MD, Principal Investigator — CHUV (Centre Hospitalier Universitaire Vaudois) Lausanne